CLINICAL TRIAL: NCT06402045
Title: Assessment of the Occlusal Characteristics and Orthodontic Treatment Needs for Egyptian Children( 6-12)Years Old
Status: Not yet recruiting | Type: Observational
Sponsor: Salma Hassan Widatalla Omar (Other)
Responsible Party: Sponsor-Investigator, Salma Hassan Widatalla Omar, principal invistigator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: ocop
Record Dates: First submitted 2024-04-30; First posted 2024-05-07 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Occlusion
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to assess the occlusal characteristics of Egyptian children 6-12 years old and their need for orthodontic treatment.

DETAILED DESCRIPTION:
The term malocclusion encompasses all deviations of teeth and jaws from normal alignment and relations including discrepancies between teeth and jaw size, malposition of individual teeth ,and mal-relationship of the dental arches in sagittal ,transverse, and vertical dimensions. The etiology of malocclusion may be due to genetic factors , environmental factors or more commonly a combination of both inherited and environmental acting together such as adverse oral habits , anomalies in number ,form ,and developmental position of teeth can cause malocclusion .The recognition of these disorders in dentistry implies the need for planning preventive ,interceptive ,and corrective orthodontic measures to provide adequate treatment .for such planning ,it is essential to carry out epidemiological studies of malocclusion prevalence and to assess the treatment need for such disorders ,so that early recognition of developing malocclusions and the potential for uncomplicated orthodontic treatment procedures can minimize or eliminate future costly treatment .

ELIGIBILITY:
Inclusion Criteria:

* Egyptian children of both genders born to Egyptian parents .
* Children having an age range from 6-12 years old.
* Cooperative children .

Exclusion Criteria:

* Craniofacial anomalies that affect jaw relation and dentition except for cleft lip and palate.
* History of facial trauma or surgery.
* Systemic disease that affects craniofacial growth
* Previously orthodontically treated child Those whom did not sign the consent

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Egyptian children of both genders born to Egyptian parents . Children having an age range from 6-12 years old.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Molar relationship (angle classification) | one year
  occlusion characteristics

SECONDARY OUTCOMES:
crowding | one year
  occlusion characteristics
Degree of overbite | one year
  occlusion characteristics
Degree of overjet | one year
  occlusion characteristics
Open bite | one year
  occlusion characteristics
Assessment of orthodontic treatment needs | one year
  occlusion characteristics
Posterior crossbite (unilateral, bilateral) | one year
  occlusion characteristics

REFERENCES:
- [Background] Alhammadi MS, Halboub E, Fayed MS, Labib A, El-Saaidi C. Global distribution of malocclusion traits: A systematic review. Dental Press J Orthod. 2018 Nov-Dec;23(6):40.e1-40.e10. doi: 10.1590/2177-6709.23.6.40.e1-10.onl. PMID 30672991
- [Background] Akbari M, Lankarani KB, Honarvar B, Tabrizi R, Mirhadi H, Moosazadeh M. Prevalence of malocclusion among Iranian children: A systematic review and meta-analysis. Dent Res J (Isfahan). 2016 Sep;13(5):387-395. doi: 10.4103/1735-3327.192269. PMID 27857763
- [Background] Nur Yilmaz RB, Oktay I, Ilhan D, Fisekcioglu E, Ozdemir F. Normative and subjective need for orthodontic treatment within different age groups in a population in Turkey. Niger J Clin Pract. 2017 Dec;20(12):1632-1638. doi: 10.4103/1119-3077.224126. PMID 29378999
- See also: cross sectional study — https://pubmed.ncbi.nlm.nih.gov/30672991/